CLINICAL TRIAL: NCT04355104
Title: Effects of Low Back Pain Knowledge-Related Education on Attitudes and Knowledge in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 810/2019
Record Dates: First submitted 2020-03-23; First posted 2020-04-21 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain
Keywords: Knowledge; Attitude; Disability; Pain
MeSH Terms: conditions — Low Back Pain; Behavior; Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education+standard physical therapy (Experimental): Consist of 37 patients will take education sessions in addition to standard physical therapy.
  Interventions: Behavioral: Education; Behavioral: Standard physical therapy
- Standard physical therapy (Active Comparator): Consist of 37 patients take just standard physical therapy.
  Interventions: Behavioral: Standard physical therapy

INTERVENTIONS:
Behavioral: Education — A one hour educational session per week for 4 weeks. In a total of 4 sessions of education, the content based on LBP Clinical Practice Guidelines which recommended that education and counseling strategies for patients with low back pain.
  Education session will be through video lecturing as a motivated tool of education for all subject who are in experimental group, this video will repeated the same in every educational session and will be sent for all participants.
  The neuroscience education will be by the therapist using interactive slide show and hand-drawing images.
  In addition to the education video, slide show, we will specify the education for every patient to give him all that he need, questions and details, mention his case on real spine to explore it and to determine the expected goal from what he need and what we have.
  Arms: Education+standard physical therapy
Behavioral: Standard physical therapy — Two session physical therapy per week for 4 weeks. The physical therapy will be based on patients case.

SUMMARY:
Low back pain (LBP) is the leading musculoskeletal condition in burden of disease and years lived with disability. This high ranking is in large part due to the high prevalence of LBP. LBP is not only mechanically related to spinal pathophysiology (i.e., postural alterations, articular stiffness, or muscle weakness), but may also be influenced by psychosocial factors such as attitudes and beliefs. Multidisciplinary rehabilitation programs, which include biopsychosocial management, resulted in a better outcome. The aim of this project is to determine if the change in LBP-related knowledge and attitudes toward LBP are correlated with the change in LBP-related pain, disability, fear avoidance, and emotional states of depression, anxiety, and stress after three months. The second aim is to investigate the effect of adding LBP knowledge related education sessions to standard physical therapy treatment on patients' LBP knowledge, attitudes toward LBP, LBP-related pain, disability, fear avoidance, and emotional symptoms in comparison to standard physical therapy alone.

DETAILED DESCRIPTION:
Low back pain (LBP) is the leading musculoskeletal condition in burden of disease and years lived with disability. This high ranking is in large part due to the high prevalence of LBP. LBP is not only mechanically related to spinal pathophysiology (i.e., postural alterations, articular stiffness, or muscle weakness), but may also be influenced by psychosocial factors such as attitudes and beliefs. Multidisciplinary rehabilitation programs, which include biopsychosocial management, resulted in a better outcome. The aim of this project is to determine if the change in LBP-related knowledge and attitudes toward LBP are correlated with the change in LBP-related pain, disability, fear avoidance, and emotional states of depression, anxiety, and stress after three months. Secondly, the investigators will investigate the effect of adding LBP knowledge related education sessions to standard physical therapy treatment on patients' LBP knowledge, attitudes toward LBP, LBP-related pain, disability, fear avoidance, and emotional symptoms in comparison to standard physical therapy alone. 74 patients with LBP receiving standard physical therapy service for the first time will be interviewed and their knowledge and attitude about LBP will be collected at the baseline. After 3 months, the LBP related pain, emotional symptoms, and LBP disability will be collected. The patients will be allocated to "Experimental group" consist of 37 patients will take education sessions in addition to standard physical therapy for 12 sessions or "control group" consist of 37 patients take just standard physical therapy for the same number of sessions without education. Participants will be assessed at baseline and at 3 months follow up. Outcome measures include Arabic version of the Back Pain Attitudes (Back-PAQ), Low Back Pain Knowledge (LKQ) Questionnaires, Arabic version of Oswestry Disability Index (ODI) to assess the function, Visual Analogue Scale for pain intensity, Depression Anxiety Stress Scales (DASS-21) for emotional states, and Fear-Avoidance Beliefs Questionnaire (FABQ) for fear avoidance beliefs. Spearman correlation coefficient r will be used to investigate the correlation between change in LBP knowledge and attitude, and change in pain, disability, fear avoidance and emotional symptoms after three months. Independent sample t-test will be used to compare the knowledge, attitude, VAS, ODI, FABQ, and DASS- between the experimental group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients reported persistent LBP of more than 3/10 in the last 12 weeks.

Exclusion Criteria:

* Subjects with acute low back pain, "red flags" indicating signs of serious pathology, previous back surgery, pregnancy, specific rheumatological diseases, spodylolysis or spondylolisthesis, spinal tumor or spinal fracture, mental disorders, or neurological diseases will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Back Pain Attitude Questionnaire from baseline to 4 weeks and 3 months | Change from baseline to 4 weeks and 3 months
  Back Pain Attitude Questionnaire is a valid, reliable instrument with acceptable internal consistency (α=0.70; 95% CI 0.66 to 0.73) used to assess beliefs about back pain among the general public, people with back pain and health professionals. It contains 34 items, divided into 6 sections with a five-point Likert scale, and response options ranging from 'False' to 'True' for each one.14 The score range from 0-34 with higher scores indicate a negative attitude toward LBP.
Change in Low Back Pain Knowledge questionnaire from baseline to 4 weeks and 3 months | Change from baseline to 4 weeks and 3 months
  Low Back Pain Knowledge questionnaire evaluates a person's knowledge of low back pain. It is a valid, reliable and sensitive to change instrument consists of 16 multiple-choice questions divided into three topics: general aspects (Questions 1, 6, 7, 8, 15), with a maximum score of nine, concepts (Questions 2, 3, 4, 5), with a maximum score of four, and treatment (Question 9, 10, 11, 12, 13, 14, 16), with a maximum score of 11. The overall maximum score of the questionnaire was 24.13 The higher score reflects a higher knowledge.
Change in Oswestry Disability Index from baseline to 4 weeks and 3 months | Change from baseline to 4 weeks and 3 months
  It measures the patient's permanent functional disability due to low back pain. It is a valid, reliable assessment tool with acceptable internal consistency (Cronbach α ranges from .71 to .87) and test-retest reliability ((r=0.83-0.99) vary according to the time interval between measurement), diagnosed to collect information about the effect of low back pain on an individual's ability to manage everyday life. Intraclass correlation coefficient values from (0.84-0.94). It includes 9 sections with a total possible score of 5 for each one. The total score which ranges from 0%-20% represents a minimal disability and from 81%-100% is represent the highest disability .
Change in Visual analogue scale from baseline to 4 weeks and 3 months | Change from baseline to 4 weeks and 3 months
  It measures the level of pain intensity. It is a valid, reliable, acceptable and sensitive to change unidimensional assessment scale of pain intensity, with acceptable (test-retest reliability (r=0.71-0.94,p<0.001)) and construct validity. The scale consists of an 11 point likert rating scale (with response options from "no pain" "0 score" to "worst pain ever" "10 score").

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales (DASS-21) from baseline to 4 weeks and 3 months | Change from baseline to 4 weeks and 3 months
  Depression Anxiety Stress Scales (DASS-21) measures the emotional states of depression, anxiety, and stress. It is a valid and reliable assessment tool, includes a set of three self-reports (7 items for each divided into subscales) with five verbal (normal, mild, moderate, severe, and extremely severe) and numeric classifications for each one, designed to measure the emotional states of depression, anxiety, and stress. (Cronbach's α = 0.94, 0.87, 0.91 for depression, anxiety and stress respectively). The higher the score in each subscale reflects higher mental symptoms.
Change in Fear-Avoidance Beliefs Questionnaire (FABQ) from baseline to 4 weeks and 3 months. | Change from baseline to 4 weeks and 3 months
  It measures the impact of patient's fear-avoidance beliefs about physical activity and work on low back pain and resulting disability. FABQ is a valid and reliable assessment questionnaire (ICC = 0.97) consist of 16 items, divided into two subscales, work (items 6, 7, 9, 10, 11, 12, 15) and physical activity (items 2, 3, 4, 5), with a maximum score of 96. A higher score reflects a higher avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Saddam F Kanaan, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No